CLINICAL TRIAL: NCT02452996
Title: A Randomised, Double-Blind, Placebo Controlled, Single Ascending Doses Study With GNbAC1 in Healthy Male Volunteers
Brief Title: Safety Study of GNbAC1 Monoclonal Antibody in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeNeuro Innovation SAS (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNC-001bis; 2014-005113-23 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2015-08

CONDITIONS: Healthy Volunteers
Keywords: GNbAC1; Multiple Sclerosis; Multiple Sclerosis Associated Retrovirus (MSRV); MSRV-Envelope protein; Monoclonal antibody; Temelimab
MeSH Terms: conditions — Multiple Sclerosis | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 6 mg/kg GNbAC1 (Active Comparator): 7 subjects randomized 5:2 active treatment:placebo
  Interventions: Drug: GNbAC1
- 18 mg/kg GNbAC1 (Active Comparator): 7 subjects randomized 5:2 active treatment:placebo
  Interventions: Drug: GNbAC1
- 36 mg/kg GNbAC1 (Active Comparator): 7 subjects randomized 5:2 active treatment:placebo
  Interventions: Drug: GNbAC1

INTERVENTIONS:
Drug: GNbAC1 — Single dose of IMP, IV infusion

SUMMARY:
In this clinical study, the safety and tolerability of GNbAC1 as a treatment for MS patients will be evaluated in healthy male volunteers.

DETAILED DESCRIPTION:
The monoclonal antibody, GNbAC1, targets the envelope protein (Env) of the human endogenous retrovirus (HERV), also called multiple sclerosis associated retrovirus (MSRV), which is considered as a critical factor in the development of multiple sclerosis.

This study will assess the pharmacokinetics, safety and tolerability of GNbAC1 following single ascending doses (6, 18, and 36 mg/kg) administered via IV infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by past medical history, physical examination, vital signs, ECG and laboratory tests at Screening and confirmed at Day -1 who have signed the informed consent.
* Aged from 18 to 55 years, both inclusive.

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of any allergy requiring acute or chronic treatment (seasonal allergic rhinitis that requires no treatment may be tolerated).
* Need of any prescription medication within 15 days prior to the administration of the study drug and/or non-prescription medication within 7 days prior to the administration of the study drug or anticipated need for any concomitant medication during the study.
* Participation in a clinical trial during the previous 3 months, i.e. from completion of the previous trial to the planned first administration of the current trial.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of single ascending doses of GNbAC1 in healthy male subjects | 57 days
  AE, SAE, vital signs, ECG, clinical laboratory values

SECONDARY OUTCOMES:
PK characteristics: GNbAC1 serum concentrations | 57 days
  GNbAC1 serum concentrations over time
immunogenicity in terms of antibodies against GNbAC1 (anti-drug antibodies) | 57 days
  antibodies against GNbAC1 (anti-drug antibodies)
ratio of serum to CSF GNbAC1 concentration | 29 days
  GNbAC1 cerebrospinal fluid concentration at Day 2 and Weeks 2 and 4 after administration

CONTACTS AND LOCATIONS:
Overall Officials: Georg Golor, MD, Principal Investigator — Parexel
Locations (1):
- PAREXEL Early Phase Clinical Unit, Berlin, Germany